CLINICAL TRIAL: NCT01054105
Title: The Prevalence of BMPR-2 Gene Mutations in Korean Patients With Pulmonary Arterial Hypertension (PAH) and the Effects of Gene Mutations on Hemodynamic Response by Drug Therapy
Brief Title: Effect of BMPR-2 Gene Mutations on Hemodynamic Response by Iloprost Inhalation in Pulmonary Arterial Hypertension
Acronym: PILGRIM
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); The Catholic University of Korea (Other); Bayer (Industry)
Responsible Party: Principal Investigator, Wook-Jin Chung, Professor, Gachon University Gil Medical Center
Other Study IDs: WJC-IIT-1001; GIRBA 2278 (Other: Gachon University Gil Hospital IRB)
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary hypertension; genes; mutation; drug therapy
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Iloprost

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BMPR-2 genes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Step I: BMPR-2 gene analysis: BMPR-2 gene analysis on 100 IPAH or heritable PAH Patients
  Interventions: Drug: Iloprost
- Step-II: Iloprost and Exercise Echo: Illoprost inhalation for 3 months & Check-up before and after treatment; WHO functional classification Assessment of exercise capacity (6M walk test) Cardiopulmonary exercise echocardiography NT-proBNP
  Interventions: Drug: Iloprost

INTERVENTIONS:
Drug: Iloprost — Iloprost inhalation, 2.5 - 5mcg, 6 times per day
  Other Names: Allowable patients from Step-I; Step-II: Illoprost and Exercise Echo

SUMMARY:
In the present study, the investigators want to investigate the prevalence of BMPR-2 gene mutations in the Korean PAH patients (Step-I) and to test that the PAH patients treated with iloprost inhalation solution (Ventavis®) would show hemodynamic response, especially assessed by exercise echocardiography (Step-II).

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) consists of a group of vascular abnormalities with elevated pulmonary arterial pressure and pulmonary vascular resistance. Idiopathic or familial PAH is progressive over several years and believed to be fatal without treatment. (1-2) The results of the Endothelin Antagonist tRial in mildly symptomatic PAH (EARLY) indicate that early diagnosis and treatment of PAH might improve time to clinical worsening and emphasize that PAH needs to be diagnosed and treated in the early stages. (3) Germline mutations of bone morphogenetic protein receptor (BMPR)-2, a member of the transforming growth factor (TGF)-β superfamily, have been found in familial and sporadic forms of idiopathic PAH,(4-6) and in appetite-suppressant PAH.(7) The BMPR-2 gene, on chromosome 2q33, has 13 exons. Exons 1-3 encode an extracellular domain, exon 4 encodes the transmembrane domain, exons 5-11 a serine/threonine kinase domain, and exons 12 and 13 a very large intracellular C-terminus of unknown function that appears to be unique to BMPR-2. (8) Mutations in familial PAH have been reported in all exons except for 5 and 13. (9) About 10-25% of sporadic cases of idiopathic PAH are thought to have BMPR-2 mutations (10) and rare cases of PAH associated with congenital heart disease, connective tissue disease and drug induced PAH were reported. (11-12) It is likely that genetic predispositions exist based on normal variations in genes that may influence the pulmonary circulation. However, the studies regarding prevalence of BMPR-2 gene mutations in Korean patients have not been performed.

In a previous study, family members of familial PAH patients showed an increased pulmonary artery systolic pressure (PASP) rise during exercise as assessed by echocardiography. (13-14) In other study, relatives of idiopathic/familial PAH patients displayed enhanced frequency of pulmonary hypertensive response during exercise and that this response is associated with mutations in the BMPR-2 gene. (15) These results suggest that asymptomatic gene carriers, in the absence of manifest pulmonary hypertension, might have enhanced PASP during exercise and more risk to develop resting pulmonary hypertension in the future compared with patients without gene mutations. Therefore, the treatment response by variable vasodilators (ex. calcium channel blockers, endothelin antagonist or prostacyclin analogues..) may be different based on the presence of BMPR-2 gene. In the present study, we want to investigate the prevalence of BMPR-2 gene mutations in the Korean PAH patients(Step-I) and to test that the PAH patients treated with iloprost inhalation solution (Ventavis®) would show hemodynamic response, especially assessed by exercise echocardiography (Step-II).

ELIGIBILITY:
Inclusion Criteria:

1. The patients aged from 20 to 80 years
2. Newly diagnosed WHO category I PAH patients: Patients who meet the following criteria within 3 months obtained by right heart catheterization (mean PAP of more than 25 mm Hg at rest and mean pulmonary arterial wedge pressure (PCWP) or left ventricular end-diastolic pressure of 15 mm Hg or less) or echocardiography (peak PAP of more than 40mmHg and mean PAP more than 30mmHg).
3. Previously diagnosed PAH patients who refractory to conventional treatment except iloprost inhalation solution (Ventavis): Patients meet the echo criteria (peak PAP of more than 40mmHg and mean PAP more than 30mmHg) who have been treated with PAH medications except iloprost inhalation solution (Ventavis) after diagnosed as WHO Group 1 PAH based on prior RHC data (above criteria) but refractory to them.
4. The patients who are able to undergo low intensity exercise test (low dose bicycle or walking)

Exclusion Criteria:

1. The patients with other left heart disease (category II in WHO classification of pulmonary hypertension); ex. Congestive HF, cardiomyopathy, significant valvular heart disease, significant arrhythmia, suspicious elevated PCWP.
2. The patients with category III,IV and V in WHO classification of pulmonary hypertension:

   * Pulmonary hypertension with lung disease and/or hypoxemia
   * Chronic obstructive pulmonary disease
   * Interstitial lung disease
   * Sleep disorder breathing
   * Alveolar hyperventilation disorders
   * Chronic exposure to high altitude
   * Developmental abnormalities
   * Pulmonary hypertension due to chronic thrombotic and/or embolic disease
   * Thromboembolic obstruction of the proximal pulmonary arteries
   * Thromboembolic obstruction of the distal pulmonary arteries
   * Non-thrombotic pulmonary embolism (e.g. tumor or parasitic)
   * Miscellaneous disorders affecting the pulmonary vasculature
   * Patients with contraindication to Ventavis;(Hypersensitive to Ventavis, High risk of bleeding, which can be increased by use of Ventavis (e.g. active peptic ulcer, trauma, intracranial hemorrhage)
   * Severe coronary disease
   * Unstable angina
   * History of Acute myocardial infarction within 6 months
   * Uncompensated heart failure not under close medical monitoring
   * Severe arrhythmia
   * Suspected pulmonary congestion
   * Cerebrovascular disease within 3 months (e.g. transient ischemic attack, stoke)
   * Pulmonary hypertension due to venous occlusive disease, valvular defect with dysfunction of cardiac muscle, which is independent of pulmonary hypertension)
   * Pregnancy
   * Women with high probability of pregnancy
   * Breast feeding
   * Renal failure (creatinine clearance: less than 30mL/min)
3. The patients concurrently using other pulmonary vasodilator (ex. Inhaled NO, endothelin antagonists) except PDE5 inhibitor
4. The patients with poor echo window which is unavailable to accept the echo data
5. The patients who cannot do any exercise
6. The patients who changes medication administered during ventavis treatment
7. The patients with allergic reaction to ventavis
8. The patients with other systemic disease (ex. Leukemia, MM, Sickle cell anemia, significant liver disease)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously diagnosed PAH
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2010-10; Primary Completion 2018-12-25 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary exercise test parameters | after 3 months active follow-up

SECONDARY OUTCOMES:
Major cardiovascular Events (cardiovascular mortality, all cause mortality, hospitalization) | After 2 years follow-up
  cardiovascular mortality, all cause mortality, hospitalization
Six-minutes walking test | After 3 months active follow-up
  min
WHO/NYHA class | After 3 months active follow-up
  WHO/NYHA class
Echo parameters | After 3 months active follow-up
  various echo parameters
NT-proBNP | After 3 months active follow-up
  NT-proBNP

CONTACTS AND LOCATIONS:
Overall Officials: Wook-Jin Chung, MD,PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (6):
- South Korea (6):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Gachon University Gil Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Catholic University Seoul Saint Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Sungkyunkwan University Seoul Samsung Hospital, Seoul

REFERENCES:
- [Derived] Jang AY, Kim BG, Kwon S, Seo J, Kim HK, Chang HJ, Chang SA, Cho GY, Rhee SJ, Jung HO, Kim KH, Seo HS, Kim KH, Shin J, Lee JS, Kim M, Lee YJ, Chung WJ. Prevalence and clinical features of bone morphogenetic protein receptor type 2 mutation in Korean idiopathic pulmonary arterial hypertension patients: The PILGRIM explorative cohort. PLoS One. 2020 Sep 23;15(9):e0238698. doi: 10.1371/journal.pone.0238698. eCollection 2020. PMID 32966279